CLINICAL TRIAL: NCT06929104
Title: Psychological Problems and Associated Factors in Patients With Thyroidectomy in Assiut University Hospitals
Brief Title: Psychological Problems in Post Thyroidectomy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad M Galal, Gehad M Galal, Assiut University
Other Study IDs: Eonpifcolpgma
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Post-Thyroidectomy Hypoparathyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergo thyroidectomy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Quality of life (QoL) refers to perceived well-being, and encompasses the evaluation of physical health, and physical, social, and psychological functioning .

The assessment of quality of life (QOL) post-thyroidectomy has gained significant attention in the medical community. Multiple studies have delved into the long-term consequences of thyroidectomy, aiming to evaluate the impact on patients' overall well-being and functional status. By examining numerous aspects, such as the physical, psychological, and social dimensions of QOL, researchers have provided valuable insights into the outcomes of thyroidectomy, hence contributing to improving patient care and enhancing their postoperative experiences.

DETAILED DESCRIPTION:
Regarding the psychological dimension of QOL, several studies have emphasized patients' emotional well-being post-thyroidectomy. Findings have demonstrated that, while many individuals experience temporary emotional disturbances related to the surgery, long-term psychological outcomes generally improve over time. In fact, the majority of patients report higher levels of self-esteem and body image post-thyroidectomy, as the removal of a diseased or abnormal thyroid gland can alleviate anxiety and distress associated with the underlying condition. However, additional research is needed to explore the specific factors contributing to these positive psychological outcomes and to identify potential interventions for those experiencing psychological distress following thyroidectomy .

Thyroidectomy is the treatment of choice in thyroid cancer patients, and the prevalence of thyroid cancer has shown a gradual increase over the past two decades. Thyroid surgery is also indicated in certain forms of benign thyroid disorder, such as nontoxic goiter and Graves' disease. Although thyroidectomy is a universal operation, few studies to date have investigated the impact of thyroidectomy on QOL .

ELIGIBILITY:
Inclusion Criteria:

* 1-Gender: both males and females 2- Post thyroidectomy patients: patients who will be planned to undergo different types of thyroidectomy for conditions such as thyroid cancer, benign thyroid disease (goiter), or hyperthyroidism (e.g., Graves' disease) and admitted as inpatients.

  3- Age Range: participants within certain age range (e.g., 18-75 years). 4-Consent: Ability to provide informed consent to participate in the study. 5-Stable Medical Condition:

Exclusion Criteria:

1. Patients who were previously diagnosed with any psychiatric diseases.
2. Medications: Use of medications that could affect outcome of the study e.g., antidepressants, corticosteroids and benzodiazepines
3. Pregnancy: Current pregnancy or breastfeeding.
4. Age: less than 18 years or more than 75 years old.
5. patients with any organ failure e.g (heart failure, end-stage renal disease requiring dialysis and liver failure) and cancers other than thyroid cancer.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergo thyroidectomy
Sampling Method: Probability Sample
Enrollment: 127 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of psychological problems e.g., depression, anxiety and fatigue in patients with post thyroidectomy surgery in Assiut University hospitals. | One year

IPD SHARING:
Plan to Share IPD: No